CLINICAL TRIAL: NCT06641089
Title: A Phase 3, Parallel-group, Randomized, Double-blind, 4-arm, Placebo-controlled, Multicenter Study With Risankizumab as Active Reference Arm, to Investigate the Efficacy and Safety of Subcutaneous Sonelokimab in Male and Female Participants Aged 18 Years and Over With Active Psoriatic Arthritis and Previous Inadequate Response or Intolerance to Tumor Necrosis Factor-α Inhibitors
Brief Title: Evaluation of Sonelokimab in Patients With Active Psoriatic Arthritis and Anti-TNFα Inadequate Response
Acronym: IZAR-2
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: MoonLake Immunotherapeutics AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: M1095-PSA-302
Record Dates: First submitted 2024-10-11; First posted 2024-10-15 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Arthritis, Psoriatic
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — sonelokimab; risankizumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- sonelokimab dose 1 with an induction regimen (Experimental): Subjects randomized to this arm will receive sonelokimab dose 1 subcutaneously (SC) as an induction regimen of 4 doses , followed by sonelokimab SC every 4 weeks (Q4W) maintenance dosing starting at Week 8.
  Interventions: Drug: Sonelokimab
- sonelokimab dose 2 with an induction regimen (Experimental): Subjects randomized to this arm will receive sonelokimab dose 2 SC as an induction regimen of 4 doses, followed by sonelokimab SC Q4W maintenance dosing starting at Week 8.
  Interventions: Drug: Sonelokimab
- Placebo (Placebo Comparator): Subjects randomized to this arm will receive placebo SC
  Interventions: Drug: Placebo
- risankizumab (Active Comparator): Subjects randomized to this arm will receive risankizumab SC
  Interventions: Drug: Risankizumab

INTERVENTIONS:
Drug: Sonelokimab — Sonelokimab
  Arms: sonelokimab dose 1 with an induction regimen; sonelokimab dose 2 with an induction regimen
Drug: Placebo — Placebo
  Arms: Placebo
Drug: Risankizumab — Active comparator
  Arms: risankizumab

SUMMARY:
This is a study to confirm the clinical efficacy and safety of sonelokimab compared with placebo in the treatment of adults with active psoriatic arthritis who have had a previous inadequate response or intolerance to anti-tumor necrosis factor (TNF)α therapy.

DETAILED DESCRIPTION:
M1095-PSA-302 is a Phase 3, parallel-group, randomized, double-blind, 4-arm, placebo-controlled, multicenter study with risankizumab as active reference arm to investigate the efficacy and safety of sonelokimab 60 mg and 120 mg versus placebo in adults with active psoriatic arthritis who have had a previous inadequate response or intolerance to anti-tumor necrosis factor (TNF)α therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be ≥18 years of age .
2. Participants have a confirmed diagnosis of psoriatic arthritis (PsA) per the 2006 Classification for Psoriatic Arthritis (CASPAR) criteria with symptoms for ≥6 months before the Screening Visit.
3. Participants have active disease (defined by a 68 tender joint count [TJC68] of ≥3 and a 66 swollen joint count [SJC66] of ≥3).
4. Participants have current active plaque psoriasis (PsO) or a dermatologist-confirmed history of plaque PsO.
5. Participants test negative for both rheumatoid factor and anti-cyclic citrullinated peptide at the Screening Visit.
6. Participants must have received 1 or more TNFα inhibitors for PsA or PsO and must have experienced an inadequate response to treatment with at least one TNFα inhibitor(s) given at an approved dose for ≥3 months or have stopped treatment due to safety/tolerability problems after ≥1 administration of a TNFα inhibitor.

Exclusion Criteria:

1. Participants with a known hypersensitivity to sonelokimab or any of its excipients.
2. Participants with a known hypersensitivity, or any contraindication, to risankizumab or any of its excipients or component of the container.
3. Participants who have a diagnosis of chronic inflammatory conditions other than PsO or PsA.
4. Participants with a diagnosis of inflammatory bowel disease.
5. Participants who have experienced a period of ≥3 consecutive weeks of unexplained diarrhea in the 24 weeks before the Baseline Visit.
6. Participants who have an established diagnosis of arthritis mutilans.
7. Previous exposure to sonelokimab.
8. Participants who have ever received biologic immunomodulating agents for PsA or PsO whether investigational or approved, except for those targeting TNFα

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2024-10-15 (Actual); Primary Completion 2027-01-15 (Estimated); Study Completion 2027-01-15 (Estimated)

PRIMARY OUTCOMES:
Response rate of participants achieving at least a 50% improvement in the American College of Rheumatology criteria (ACR50) | Week 16 compared to placebo
  Proportion of participants achieving ACR50

SECONDARY OUTCOMES:
Response rate of participants achieving at least 20% improvement in the American College of Rheumatology criteria (ACR20) | Week 16 compared to placebo
  Proportion of participants achieving ACR20
Response rate of participants achieving Minimal Disease Activity (MDA) | Week 16 compared to placebo
  Proportion of participants achieving MDA
Health Assessment Questionnaire- Disability Index (HAQ-DI) | Week 16 compared to placebo
  Change in HAQ-DI from baseline
Psoriasis Area and Severity Index (PASI90) | Week 16 compared to placebo
  Proportion of participants achieving a decrease of ≥90% in the PASI90 response at Week 16 in the subgroup of participants with psoriasis (PsO) involving ≥3% body surface area at baseline
Short- form-36 (SF-36) Physical Component Summary (PCS) | Week 16 compared to placebo
  Change from Baseline in SF-36 PCS at Week 16
Response rate of participants achieving at least a 50% improvement in the American College of Rheumatology criteria (ACR50) | Week 16 compared to risankzumab
  Proportion of participants achieving ACR50

CONTACTS AND LOCATIONS:
Locations (98):
- United States (43):
  - Clinical Site, Avondale, Arizona
  - Clinical Site, Chandler, Arizona
  - Clinical Site, Flagstaff, Arizona
  - Clinical Site, Mesa, Arizona
  - Clinical Site, Phoenix, Arizona
  - Clinical Site, Scottsdale, Arizona
  - Clinical Site, Tucson, Arizona
  - Clinical Site, Jonesboro, Arkansas
  - Clinical Site, Pomona, California
  - Clinical Site, San Diego, California
  - Clinical Site, Santa Monica, California
  - Clinical Site, Thousand Oaks, California
  - Clinical Site, Upland, California
  - Clinical Site, Avon Park, Florida
  - Clinical Site, Clearwater, Florida
  - Clinical Site, Hialeah, Florida
  - Clinical Site, Miami Gardens, Florida
  - Clinical Site, Tampa, Florida
  - Clinical Site, Zephyrhills, Florida
  - Clinical Site, Gainesville, Georgia
  - Clinical Site, Springfield, Illinois
  - Clinical Site, Lake Charles, Louisiana
  - Clinical Site, Baltimore, Maryland
  - Clinical Site, Grand Blanc, Michigan
  - Clinical Site, Brooklyn, New York
  - Clinical Site, Rochester, New York
  - Clinical Site, Charlotte, North Carolina
  - Clinical Site, Leland, North Carolina
  - Clinical Site, Middleburg Heights, Ohio
  - Clinical Site, Portland, Oregon
  - Clinical Site, Duncansville, Pennsylvania
  - Clinical Site, Jackson, Tennessee
  - Clinical Site, Memphis, Tennessee
  - Clinical Site, Murfreesboro, Tennessee
  - Clinical Site, Allen, Texas
  - Clinical Site, Austin, Texas
  - Clinical Site, Baytown, Texas
  - Clinical Site, Colleyville, Texas
  - Clinical Site, Houston, Texas
  - Clinical Site, Lubbock, Texas
  - Clinical Site, Plano, Texas
  - Clinical Site, Seattle, Washington
  - Clinical Site, Beckley, West Virginia
- Bulgaria (5):
  - Clinical Site, Pleven
  - Clinical Site, Plovdiv
  - Clinical Site, Rousse
  - Clinical Site, Sofia
  - Clinical Site, Stara Zagora
- Canada (5):
  - Clinical Site, Toronto, Ontario
  - Clinical Site, Calgary
  - Clinical Site, Trois-Rivières
  - Clinical Site, Waterloo
  - Clinical Site, Winnipeg
- Czechia (4):
  - Clinical Site, Brno
  - Clinical Site, Ostrava
  - Clinical Site, Studénka
  - Clinical Site, Zlín
- France (6):
  - Clinical Site, Caluire-et-Cuire
  - Clinical Site, Montpellier
  - Clinical Site, Narbonne
  - Clinical Site, Nice
  - Clinical Site, Rouen
  - Clinical Site, Tours
- Clinical Site, Tbilisi, Georgia
- Germany (6):
  - Clinical Site, Berlin
  - Clinical Site, Erlangen
  - Clinical Site, Hamburg
  - Clinical Site, Herne
  - Clinical Site, Munich
  - Clinical Site, München
- Hungary (7):
  - Clinical Site, Budapest
  - Clinical Site, Debrecen
  - Clinical SIte, Gyula
  - Clinical Site, Hódmezővásárhely
  - Clinical Site, Nyíregyháza
  - Clinical Site, Székesfehérvár
  - Clinical Site, Veszprém
- Poland (12):
  - Clinical Site, Bialystok
  - Clinical Site, Bydgoszcz
  - Clinical Site, Częstochowa
  - Clinical Site, Elblag
  - Clinical Site, Krakow
  - Clinical Site, Nadarzyn
  - Clinical Site, Poznan
  - Clinical Site, Sochaczew
  - Clinical Site, Swidnica
  - Clinical Site, Warsaw
  - Clinical Site, Wołomin
  - Clinical Site, Wroclaw
- Spain (6):
  - Clinical Site, A Coruña
  - Clinical Site, Castellon
  - Clinical Site, Madrid
  - Clinical SIte, Sabadell
  - Clinical Site, Santiago de Compostela
  - Clinical Site, Seville
- United Kingdom (3):
  - Clinical Site, Westcliff-on-Sea, Essex
  - Clinical Site, Barnet
  - Clinical Site, Leeds